CLINICAL TRIAL: NCT05042986
Title: A Phase I, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-SKI-O-703 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study of the Absorption, Metabolism, and Excretion of [14C]-SKI-O-703 Following a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OCSO-P1204
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Dose Capsule (Experimental): Single oral dose of 200 mg (100 μCi in 200 mg salt [0.5 μCi/mg as salt], equivalent to 100 μCi in 142 mg active [0.7 μCi/mg as active]) of [14C]-SKI-O-703 containing approximately 100 μCi of [14C]-SKI-O-703 per capsule after an overnight fast.
  Interventions: Drug: .[14C]-SKI-O-703

INTERVENTIONS:
Drug: .[14C]-SKI-O-703 — Single oral dose of 200 mg (100 μCi in 200 mg salt [0.5 μCi/mg as salt], equivalent to 100 μCi in 142 mg active [0.7 μCi/mg as active]) of [14C]-SKI-O-703 containing approximately 100 μCi of [14C]-SKI-O-703 per capsule after an overnight fast.

SUMMARY:
This will be a Phase I, open-label, nonrandomized, single dose study in healthy male subjects.

Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the dose administration. Subjects will be admitted into the study site on Day -1 and be confined to the study site until at least Day 8. On the morning of Day 1, all subjects will receive a single oral dose of [14C]-SKI-O-703. Subjects will be discharged if the following discharge criteria are met: plasma radioactivity levels below the limit of quantitation for 2 consecutive collections, ≥ 90% mass balance recovery, and ≤ 1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 2 consecutive 24-hour periods. If discharge criteria are not met by Day 8, subjects will remain in the study site up to Day 15.

DETAILED DESCRIPTION:
SKI-O-703 is being developed by Oscotec Inc. and is currently being studied for the treatment of adult patients with moderately to severely active rheumatoid arthritis and for the treatment of patients with persistent and chronic immune thrombocytopenia. SKI-O-592 (the free base of SKI-O-703) has demonstrated high selectivity and potency against spleen tyrosine kinase in a biochemical assay. For immunoreceptor activation linked to SYK, the effect of SKI-O-592 on the anti-inflammatory response consisting of tumor necrosis factor alpha, β-hexosaminidase, and CD69 expression was greater than the effects of first-generation SYK inhibitors (eg, R406) in several immune cell lines and in human primary cells. This anti-inflammatory activity was responsible for the selective inhibition of p-SYK (Y525/526), which led to the sequential inhibition of downstream effectors. In vitro studies revealed excellent SYK selectivity of SKI-O-592 that led to no inhibition of SYK-independent signal pathways, indicating that SKI-O-592 shows more potent anti-inflammatory activity to allow continuous administration of SKI-O-703 compared with the first-generation SYK inhibitors. SKI-O-703 is currently not approved or marketed in any country.

ELIGIBILITY:
Inclusion Criteria:

* Males, of any race, between 18 and 55 years of age, inclusive.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and/or check-in as assessed by the investigator (or designee).
* Subjects will agree to use contraception as detailed in the protocol
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
* History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). Cholecystectomy is not allowed.
* History of alcoholism or drug/chemical abuse within 2 years prior to check-in.
* Alcohol consumption of > 21 units per week. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
* Positive urine drug screen at screening or positive alcohol urine test result or positive urine drug screen at check-in.
* Positive hepatitis panel and/or positive human immunodeficiency virus test (Appendix 2).
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 5 half-lives of the drug, if known, or 30 days, whichever is longer, prior to last dose of the previous study.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, cytochrome P450 1A2 and UGT1A1 inhibitors/inducers, or elimination processes, including St. John's wort, within 30 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any prescription medications/products within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to check-in, unless deemed acceptable by the investigator (or designee).
* Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine at screening or check-in.
* Receipt of blood products within 2 months prior to check-in.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
* Poor peripheral venous access.
* Have previously completed or withdrawn from this study or any other study investigating SKI-O-703, and have previously received SKI-O-703.
* Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
* Subjects who have participated in more than 3 radiolabeled drug studies in the last 12 months (previous study to be at least 4 months prior to check-in to the study site where exposures are known to the investigator or 6 months prior to check-in to the study site for a radiolabeled drug study where exposures are not known to the investigator). The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the Code of Federal Regulations (CFR) recommended levels considered safe, per United States Title 21 CFR 361.1.5
* Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
AUC (Area under creative curve) from time zero to infinity (AUC0-∞) | Baseline through day 43
AUC from time zero to the last quantifiable concentration (AUC0-tlast) | Baseline through day 43
Time to Cmax | Baseline through day 43
Time to tmax | Baseline through day 43
Time to t1/2 | Baseline through day 43
Apparent total clearance (CL/F; plasma SKI-O-592 only) | Baseline through day 43
Apparent volume of distribution (Vz/F; plasma SKI-O-592 only) | Baseline through day 43
AUC0-∞ of plasma SKI-O-592 relative to AUC0-∞ of plasma total radioactivity (AUC0-∞ Plasma SKI-O-592/Total Radioactivity Ratio) | Baseline through day 43
AUC0-∞ of whole blood total radioactivity to AUC0-∞ of plasma total radioactivity (AUC0-∞ Blood/Plasma Ratio | Baseline through day 43
Amount of SKI-O-592 and total radioactivity excreted in urine (Aeu) | Baseline through day 43
Cumulative Aeu of SKI-O-592 and total radioactivity | Baseline through day 43
Percentage of SKI-O-592 excreted in urine (feu) and total radioactivity | Baseline through day 43
Cumulative feu of SKI-O-592 and total radioactivity | Baseline through day 43
Renal clearance (CLR; SKI-O-592 only) | Baseline through day 43
Amount of total radioactivity excreted in feces (Aef) | Baseline through day 43
Cumulative radioactivity Aef | Baseline through day 43
Percentage of total radioactivity excreted in feces (fef) | Baseline through day 43
Cumulative radioactivity fef | Baseline through day 43

SECONDARY OUTCOMES:
Metabolic profile of SKI-O-592 | Baseline through day 43
Identifications of SKI-O-592 metabolites | Baseline through day 43
Number and severity of AEs | Screening through day 43
incidence of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results | Screening through day 43
Incidence of abnormal 12-Lead ECG | Screening through day 43
Incidence of abnormal vital sign measurements | Screening through day 43
Incidence of abnormal physical examination | Screening through day 43

CONTACTS AND LOCATIONS:
Overall Officials: Study Chair, Study Chair — Oscotec Inc.
Locations (1):
- Labcorp Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No